CLINICAL TRIAL: NCT03712124
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Pilot Study of CNSA-001 in Women With Moderate to Severe Diabetic Gastroparesis
Brief Title: A Study of CNSA-001 in Women With Diabetic Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAS-001
Record Dates: First submitted 2018-10-15; First posted 2018-10-19 (Actual); Results first posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — sepiapterin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CNSA-001 (Experimental): Participants will receive CNSA-001 20 mg/kg/day (10 mg/kg twice daily [BID]) as an oral suspension for 14 days.
  Interventions: Drug: CNSA-001
- Placebo (Placebo Comparator): Participants will receive placebo matching to CNSA-001 BID for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNSA-001 — CNSA-001 Powder for Suspension
  Other Names: sepiapterin
  Arms: CNSA-001
Drug: Placebo — Placebo Suspension
  Arms: Placebo

SUMMARY:
This study evaluates CNSA-001 (sepiapterin) in the treatment of women with moderate to severe diabetic gastroparesis. Participants will be randomized in a ratio of 1:1 to receive CNSA-001 20 (milligrams) mg/kilogram (kg)/day or placebo. All participants will receive the standard of care for diabetic gastroparesis.

DETAILED DESCRIPTION:
Nerves throughout the luminal gastrointestinal (GI) tract express neuronal nitric oxide synthase (nNOS), which generates nitric oxide (NO), a key neurotransmitter in the regulation of GI motility. Several co-factors are known to be important for nNOS activity, including nicotinamide adenine dinucleotide phosphate hydrogen (NADPH), calcium, and tetrahydrobiopterin (BH4). The homodimeric conformation of all 3 isoforms of nitric oxide synthase (NOS) is regulated by BH4. In the absence of BH4, uncoupling of NO production occurs and leads to super oxide production, resulting in further impaired nNOS bioactivity.

CNSA-001 is a new chemical entity that is an endogenous, naturally occurring precursor of BH4 via the pterin salvage pathway. Oral administration of CNSA-001 will result in increases in both intracellular and circulating BH4 concentrations. Increased BH4 concentration is hypothesized to improve nNOS function resulting in a positive effect on gastric accommodation and emptying.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Diagnosis of diabetes mellitus
* Documentation of delayed gastric emptying on gastric emptying scintigraphy or gastric emptying breath test (GEBT) (within 2 year of enrollment)
* Symptoms of gastroparesis for at least 6 months with GCSI score >21 indicating moderate to severe symptoms
* Gastric accommodation, as measured by nutrient satiety testing, of ≤600 mL
* Negative upper endoscopy or upper GI series within 3 years of enrollment (no evidence of mechanical obstruction or peptic ulcer disease)
* Either postmenopausal for ≥1 year or surgically sterile (having undergone tubal ligation, hysterectomy, or bilateral oophorectomy) for at least 6 months or, if of childbearing potential and not abstinent, willing to use a highly effective method of contraception throughout the study such as 1 of the following:

  * Hormonal contraception (stable dose for 3 months)
  * Intrauterine device/Intrauterine Hormone-releasing System
  * Barrier contraceptive method (diaphragm, cervical cap, contraceptive sponge, condom)

Participants who are abstinent will not be required to use a contraceptive method unless they become sexually active.

* If on analgesics (including narcotics), promotility agents (including metoclopramide), or neuromodulators (including tricyclic antidepressants, gabapentin, and pregabalin), doses are stable for >30 days before randomization and the participant is not expected to require dose changes during the study through the end of treatment (EOT)
* Have not used tobacco (for example, cigarettes, e-cigarettes, cigars, smokeless tobacco, nicotine replacement) for 2 weeks prior to Day 1 and willingness to abstain from these products during the study through the EOT

Exclusion Criteria:

* Male gender
* Normal gastric emptying
* Gastroparesis from postsurgical etiologies
* Another active disorder that could, in the opinion of the investigator, explain symptoms
* Weight >100 kg
* Alanine aminotransferase > 2× upper limit of normal (ULN)
* Pregnant, breastfeeding, or considering pregnancy
* Clinically significant cardiac arrhythmia at screening
* QT interval corrected for heart rate (QTc) ≥470 milliseconds (msec) using Fridericia's correction (based on triplicate measurements taken at screening)
* Resting heart rate ≤40 or ≥110 beats per minute (bpm) or resting blood pressure <90/40 millimeters of mercury (mmHg) or >150/90 mmHg at screening or prior to the first administration of study drug
* Recent clinically significant GI bleeding
* Taking levodopa or domperidone within 30 days before randomization or expected to require domperidone during the study through the EOT
* Taking erythromycin within 30 days before randomization or expected to require erythromycin within 30 days before randomization or expected to require erythromycin during the study; if a participant is taking erythromycin and is otherwise eligible to participate in the study, following informed consent, the participant may go through an erythromycin washout period of 30 days before randomization
* Taking any fundic-relaxing agents including, but not limited to, buspirone, clonidine, nitrates, phosphodiesterase inhibitors (that is, sildenafil citrate [Viagra®]) and triptan containing medications, within 30 days before randomization or expected to require any of these agents during the study through the EOT
* Taking any systemic antifolates, including, but not limited to, methotrexate, pemetrexed, and trimetrexate or expected to require any systemic antifolates during the study (topical antifolates [for example, cream, ointment, gel] or eye drops with antifolates are allowed)
* Pulmonary dysfunction (for example, chronic obstructive pulmonary disease)
* Surgery for placement of a gastric stimulator within the past 6 months (participants postoperative >6 months with persistent symptoms and delayed gastric emptying are eligible)
* Gastrointestinal disease (such as irritable bowel syndrome, inflammatory bowel disease, chronic gastritis, peptic ulcer disease, small bowel malabsorption) that could affect the absorption of study drug or contraindicate undergoing the GEBT
* History of gastric surgery, including Roux-en-Y gastric bypass surgery or an antrectomy with vagotomy, or gastrectomy
* History of allergies or adverse reactions to BH4 or related compounds, to any excipients in the study drug formulation, or to egg, wheat, or algae (Spirulina)
* Inability to tolerate oral medication
* Current participation in any other investigational drug study or use of any investigational agent, investigational device, or approved therapy for investigational use within 30 days or 5 half lives (whichever is longer) before screening
* Any clinically significant laboratory abnormality; in general, each laboratory value from screening and baseline chemistry and hematology panels should fall within the limits of the normal laboratory reference range unless deemed not clinically significant by the investigator
* Major surgery within the previous 90 days
* The participant, in the opinion of the investigator, is unwilling or unable to adhere to the requirements of the study
* History of alcohol or drug abuse within 6 months prior to screening or current evidence of substance dependence as determined by the investigator
* Episodes of ketoacidosis or hypoglycemia that are frequent as defined by the investigator
* History of phenylketonuria (PKU) or hyperphenylalaninemia
* Any other conditions, including diabetic comorbidities, that, in the opinion of the investigator or sponsor, would interfere with the participant's ability to participate in the study or increase the risk of participation for that participant

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-09-08 (Actual); Study Completion 2019-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Smith, PharmD, Study Director — Censa Pharmaceuticals
Locations (6):
- United States (6):
  - GW Research, Inc., Chula Vista, California
  - LMG Research, Miami, Florida
  - Indiana University Hospital, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Clinical Research Solutions, LLC, Jackson, Tennessee

REFERENCES:
- [Derived] Abell TL, Garcia LM, Wiener GJ, Wo JM, Bulat RS, Smith N. Effect of Oral CNSA-001 (sepiapterin, PTC923) on gastric accommodation in women with diabetic gastroparesis: A randomized, placebo-controlled, Phase 2 trial. J Diabetes Complications. 2021 Sep;35(9):107961. doi: 10.1016/j.jdiacomp.2021.107961. Epub 2021 Jun 17. PMID 34176722

RESULTS

PARTICIPANT FLOW:
Groups:
- CNSA-001: Participants received CNSA-001 (sepiapterin) 20 milligrams (mg)/kilogram (kg)/day (10 mg/kg twice daily [BID]) as an oral suspension for 14 days.
- Placebo: Participants received placebo matched to CNSA-001 BID for 14 days.
Period: Overall Study
Arm/Group | CNSA-001 | Placebo
Started | 10 | 11
Received at Least 1 Dose of Study Drug | 10 | 11
Completed | 9 | 11
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any amount of study drug (CNSA-001 or placebo).
Groups:
- CNSA-001: Participants received CNSA-001 20 mg/kg/day (10 mg/kg BID) as an oral suspension for 14 days.
- Total: Total of all reporting groups
Arm/Group | CNSA-001 | Placebo | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (14.29) | 60.5 (15.53) | 54.4 (15.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 10 | 15
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Day 1) in Maximal Tolerated Volume Consumed During the Nutrient Satiety Test at Day 14
Description: Participants consumed 150 milliliters (mL) of Ensure™ every 5 minutes for the nutrient satiety test. At 5-minute intervals, participants scored their fullness using a rating scale that combines verbal descriptors on a scale graded 0 to 5 (0 = no symptoms, 1 = first sensation of fullness [threshold], 2 = mild, 3 = moderate, 4 = severe and 5 = maximum or unbearable fullness). Participants were told to stop when a score of 5 was obtained. The actual volume of Ensure™ consumed at this point was the maximum tolerated volume.
Time Frame: Baseline (Day 1), Day 14
Population: Safety population included all participants who received any amount of study drug (CNSA-001 or placebo). Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | CNSA-001 | Placebo
Number analyzed (Participants) | 10 | 11
mL
  Baseline | 293.5 (124.52) | 345.6 (99.06)
  Change at Day 14: number analyzed (Participants) | 9 | 11
  Change at Day 14 | 1.3 (145.51) | 2.0 (72.61)
Statistical Analysis 1: Comparison: CNSA-001 vs Placebo; Analysis was performed using an analysis of covariance (ANCOVA) model with change from baseline at Day 14 as the dependent variable and baseline maximum tolerated volume and treatment as covariates; Test type: Other; p = 0.9030, ANCOVA; Least Square (LS) Mean Difference = -6.44, 95% CI 2-sided [-116.18 to 103.31]

2. Primary Outcome: Change From Baseline (Day 1) in Maximal Tolerated Volume Consumed During the Nutrient Satiety Test at Day 28
Description: Participants consumed 150 mL of Ensure™ every 5 minutes for the nutrient satiety test. At 5-minute intervals, participants scored their fullness using a rating scale that combines verbal descriptors on a scale graded 0 to 5 (0: no symptoms, 1 = first sensation of fullness [threshold], 2 = mild, 3 = moderate, 4 = severe and 5 = maximum or unbearable fullness). Participants were told to stop when a score of 5 was obtained. The actual volume of Ensure™ consumed at this point was the maximum tolerated volume.
Time Frame: Baseline (Day 1), Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | CNSA-001 | Placebo
Number analyzed (Participants) | 10 | 11
mL
  Baseline | 293.5 (124.52) | 345.6 (99.06)
  Change at Day 28: number analyzed (Participants) | 8 | 11
  Change at Day 28 | 75.3 (61.40) | -30.9 (67.00)
Statistical Analysis 1: Comparison: CNSA-001 vs Placebo; Analysis was performed using ANCOVA model with change from baseline at Day 28 as the dependent variable and baseline maximum tolerated volume and treatment as covariates; Test type: Other; p = 0.0042, ANCOVA; LS Mean Difference = 98.45, 95% CI 2-sided [35.81 to 161.08]

3. Secondary Outcome: Change From Baseline (Day 1) in the Gastroparesis Cardinal Symptom Index (GCSI) Total Score at Day 14/15 and Day 28
Description: The GCSI consists of 9 symptom severity items covering the following domains (subscales): nausea/vomiting (Questions 1 to 3); post-prandial fullness/early satiety (Questions 4 to 7), and bloating (Questions 8 and 9). Each question was rated on a 6-point Likert scale (0 = None, 1 = Very Mild, 2 = Mild, 3 = Moderate, 4 = Severe and 5 = Very Severe), with lower scores representing lesser symptom severity. To obtain a participant-specific score on each subscale, the scores on each question within the subscale were summed for each participant and divided by the number of questions in the subscale. Total GCSI score was mean of 3 subscales. Total aggregate GCSI score ranges from 0 to 45, with lower scores indicating lesser symptom severity.
Time Frame: Baseline (Day 1), Days 14/15 and 28
Population: Safety population included all participants who received any amount of study drug (CNSA-001 or placebo). Here, 'Number analyzed' signifies participants evaluable for this outcome measure for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CNSA-001 | Placebo
Number analyzed (Participants) | 10 | 11
units on a scale
  Baseline | 3.1778 (0.78951) | 3.3030 (0.68329)
  Change at Day 14/15: number analyzed (Participants) | 9 | 11
  Change at Day 14/15 | -1.0864 (0.82921) | -1.0101 (0.94602)
  Change at Day 28: number analyzed (Participants) | 8 | 11
  Change at Day 28 | -0.9583 (1.12677) | -0.8081 (0.98519)

4. Secondary Outcome: Change From Baseline (Day 1) in the Patient Assessment of Upper Gastrointestinal Disorders-Symptom Severity (PAGI-SYM) Subscale Scores at Day 14 and Day 28
Description: The PAGI-SYM is a 20-item upper gastrointestinal (GI) symptom severity instrument with 6 subscales: nausea/vomiting (Questions 1 to 3), post-prandial fullness/early satiety (Questions 4 to 7), bloating (Questions 8 and 9), upper abdominal pain (Questions 10 and 11), lower abdominal pain (Questions 12 and 13), and heartburn/regurgitation (Questions 14 to 20). Each question was rated on a 6-point Likert scale (0 = None, 1 = Very Mild, 2 = Mild, 3 = Moderate, 4 = Severe and 5 = Very Severe), with lower scores representing lesser symptom severity. To obtain a participant-specific score on each subscale and the total PAGI-SYM, the scores on each question within the subscale were summed for each participant and divided by the number of questions in the subscale.
Time Frame: Baseline (Day 1), Days 14 and 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CNSA-001 | Placebo
Number analyzed (Participants) | 10 | 11
units on a scale
  Nausea/Vomiting Subscale Score: Baseline | 1.7667 (1.25757) | 1.7879 (1.19511)
  Nausea/Vomiting Subscale Score: Change at Day 14: number analyzed (Participants) | 9 | 11
  Nausea/Vomiting Subscale Score: Change at Day 14 | -0.4074 (0.64070) | -0.6970 (0.88763)
  Nausea/Vomiting Subscale Score: Change at Day 28: number analyzed (Participants) | 8 | 11
  Nausea/Vomiting Subscale Score: Change at Day 28 | -0.2500 (0.72921) | -0.7273 (1.31503)
  Fullness Subscale Score: Baseline | 4.025 (0.9461) | 4.068 (0.7753)
  Fullness Subscale Score: Change at Day 14: number analyzed (Participants) | 9 | 11
  Fullness Subscale Score: Change at Day 14 | -1.278 (1.1622) | -1.023 (1.1750)
  Fullness Subscale Score: Change at Day 28: number analyzed (Participants) | 8 | 11
  Fullness Subscale Score: Change at Day 28 | -1.344 (1.6687) | -0.818 (1.2554)
  Bloating Subscale Score: Baseline | 4.25 (0.979) | 4.09 (1.020)
  Bloating Subscale Score: Change at Day 14: number analyzed (Participants) | 9 | 11
  Bloating Subscale Score: Change at Day 14 | -1.67 (0.612) | -1.23 (1.348)
  Bloating Subscale Score: Change at Day 28: number analyzed (Participants) | 8 | 11
  Bloating Subscale Score: Change at Day 28 | -1.69 (1.361) | -1.05 (1.036)
  Upper Abdominal Pain Subscale Score: Baseline | 2.55 (1.343) | 3.00 (0.975)
  Upper Abdominal Pain Score: Change at Day 14: number analyzed (Participants) | 9 | 11
  Upper Abdominal Pain Score: Change at Day 14 | -0.94 (0.917) | -1.00 (1.360)
  Upper Abdominal Pain Score: Change at Day 28: number analyzed (Participants) | 8 | 11
  Upper Abdominal Pain Score: Change at Day 28 | -0.69 (1.413) | -1.00 (1.323)
  Lower Abdominal Pain Subscale Score: Baseline | 2.20 (1.337) | 2.41 (1.429)
  Lower Abdominal Pain Score: Change at Day 14: number analyzed (Participants) | 9 | 11
  Lower Abdominal Pain Score: Change at Day 14 | -0.39 (0.821) | -0.68 (1.383)
  Lower Abdominal Pain Score: Change at Day 28: number analyzed (Participants) | 8 | 11
  Lower Abdominal Pain Score: Change at Day 28 | -0.19 (1.668) | -0.23 (1.126)
  Heartburn Subscale Score: Baseline | 2.3571 (0.84448) | 2.7013 (1.39453)
  Heartburn Subscale Score: Change at Day 14: number analyzed (Participants) | 9 | 11
  Heartburn Subscale Score: Change at Day 14 | -0.9048 (1.08327) | -1.0260 (1.23357)
  Heartburn Subscale Score: Change at Day 28: number analyzed (Participants) | 8 | 11
  Heartburn Subscale Score: Change at Day 28 | -0.7143 (1.26629) | -0.7922 (0.55462)

5. Secondary Outcome: Change Form Baseline (Day 1) in the Gastric Emptying Breath Test (GEBT) Excretion Rate at Day 14 and Day 28
Description: The GEBT is a nonradioactive non-invasive test, conducted over a 4-hour evaluation period and is designed to show how rapidly the stomach empties solids by measuring carbon dioxide (CO2) in a participant's breath. The GEBT measures the rate of CO2 excretion after consumption of a C-enriched test meal. The participant's CO2 excretion rate at any measurement time "t" was calculated and reported using the GEBT metric "kPCD". kPCD stands for "1000 * Percent Carbon-13 Dose (PCD) excreted per minute." Participants provided baseline (premeal) breath samples and then consumed a standardized 230 kilocalorie (kCal) meal. Single post-meal breath samples were collected in capped glass tubes at 45, 90, 120, 150, 180, and 240 minutes after the meal was consumed. The GEBT kPCD value (13CO2 excretion rate) was proportional to the rate of gastric emptying. Increasing GEBT values represent increasing rates of gastric emptying.
Time Frame: Baseline (Day 1), Days 14 and 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kPCD
Arm/Group | CNSA-001 | Placebo
Number analyzed (Participants) | 10 | 11
kPCD
  Baseline: 45 minutes post-meal | 5.85 (3.727) | 9.45 (3.125)
  Baseline: 90 minutes post-meal | 14.62 (8.697) | 16.10 (5.414)
  Baseline: 120 minutes post-meal | 22.59 (12.859) | 22.96 (7.139)
  Baseline: 150 minutes post-meal | 28.13 (15.552) | 28.75 (8.257)
  Baseline: 180 minutes post-meal | 31.87 (17.553) | 32.80 (9.733)
  Baseline: 240 minutes post-meal | 34.50 (17.129) | 37.32 (10.854)
  Change at Day 14: 45 minutes post-meal: number analyzed (Participants) | 9 | 11
  Change at Day 14: 45 minutes post-meal | 5.68 (7.984) | 1.55 (4.954)
  Change at Day 14: 90 minutes post-meal: number analyzed (Participants) | 9 | 11
  Change at Day 14: 90 minutes post-meal | 7.33 (12.049) | 1.67 (3.914)
  Change at Day 14: 120 minutes post-meal: number analyzed (Participants) | 9 | 11
  Change at Day 14: 120 minutes post-meal | 7.03 (15.646) | 2.14 (6.549)
  Change at Day 14: 150 minutes post-meal: number analyzed (Participants) | 9 | 11
  Change at Day 14: 150 minutes post-meal | 5.60 (16.822) | 2.02 (8.163)
  Change at Day 14: 180 minutes post-meal: number analyzed (Participants) | 9 | 11
  Change at Day 14: 180 minutes post-meal | 4.71 (19.282) | 3.34 (7.294)
  Change at Day 14: 240 minutes post-meal: number analyzed (Participants) | 9 | 11
  Change at Day 14: 240 minutes post-meal | 0.67 (19.535) | 1.18 (10.426)
  Change at Day 28: 45 minutes post-meal: number analyzed (Participants) | 8 | 11
  Change at Day 28: 45 minutes post-meal | 2.28 (5.109) | 2.00 (3.326)
  Change at Day 28: 90 minutes post-meal: number analyzed (Participants) | 8 | 11
  Change at Day 28: 90 minutes post-meal | 0.76 (11.739) | 4.42 (8.625)
  Change at Day 28: 120 minutes post-meal: number analyzed (Participants) | 8 | 11
  Change at Day 28: 120 minutes post-meal | 0.26 (13.656) | 3.59 (11.081)
  Change at Day 28: 150 minutes post-meal: number analyzed (Participants) | 8 | 11
  Change at Day 28: 150 minutes post-meal | -0.34 (14.750) | 2.39 (9.609)
  Change at Day 28: 180 minutes post-meal: number analyzed (Participants) | 8 | 11
  Change at Day 28: 180 minutes post-meal | 0.44 (11.714) | 1.43 (9.221)
  Change at Day 28: 240 minutes post-meal: number analyzed (Participants) | 8 | 11
  Change at Day 28: 240 minutes post-meal | 0.43 (11.656) | -1.43 (9.286)

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline up to Day 44
Population: Safety population included all participants who received any amount of study drug (CNSA-001 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | CNSA-001 | Placebo
Number analyzed (Participants) | 10 | 11
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: Baseline up to Day 44
Description: Safety population included all participants who received any amount of study drug (CNSA-001 or placebo).
Arm/Group | CNSA-001 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/10 | 0/11
Other Adverse Events (participants affected / at risk) | 2/10 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CNSA-001 (N=10) | Placebo (N=11)
Impaired gastric emptying (Gastrointestinal disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CNSA-001 (N=10) | Placebo (N=11)
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT03712124/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT03712124/SAP_001.pdf